CLINICAL TRIAL: NCT04795167
Title: FlowTriever for Acute Massive Pulmonary Embolism (FLAME)
Acronym: FLAME
Status: Completed | Type: Observational
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-001
Record Dates: First submitted 2021-03-04; First posted 2021-03-12 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: PE - Pulmonary Embolism; PE - Pulmonary Thromboembolism
Keywords: PE; pulmonary embolism; thromboembolism; thrombectomy; FlowTriever; massive pulmonary embolism; high risk pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FlowTriever Arm: FlowTriever Arm subjects are defined as those subjects where FlowTriever is used as the Primary Treatment for pulmonary embolism.
- Context Arm: Subjects with high-risk pulmonary embolism who are treated with non-FlowTriever therapies.
- Prior Therapy Arm: Subjects presenting with low/intermediate-risk PE who received advanced therapy but subsequently progressed to high-risk PE in the same hospital setting/admission.

SUMMARY:
To evaluate treatment outcomes of patients diagnosed with high-risk (massive) pulmonary embolism

ELIGIBILITY:
Inclusion Criteria:

Age >=18 years Treatment team determines pulmonary embolism is the cause of shock, and the PE is high-risk per the protocol definitions

Exclusion Criteria:

* Out of hospital cardiac arrest with Glasgow Coma Scale of ≤8
* Witnessed cardiac arrest with ongoing CPR >30 minutes
* Contraindication to anticoagulants, i.e. heparin or alternative
* Hematocrit <28%
* Platelets <25,000/μL
* INR >8
* Intracardiac thrombus and/or intracardiac clot in transit
* Known anaphylactic sensitivity to radiographic agents that cannot be pre-treated
* History of pulmonary hypertension with systolic pulmonary arterial pressure >70 mmHg
* Presence of chronic medical conditions with estimated < 90 days life expectancy per physician discretion (should not consider the current pulmonary embolism and its treatment)
* Current participation in another drug or device treatment study that, in the Investigator's opinion, would interfere with participation in this study
* Patient is known to be COVID-19 positive at hospital admission (patient has active COVID-19)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk (massive) pulmonary embolism.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Silver, MD, Principal Investigator — OhioHealth Riverside; James Horowitz, MD, Principal Investigator — NYU Langone Medical Center
Locations (11):
- United States (11):
  - Emory University, Atlanta, Georgia
  - Beaumont Royal Oak, Royal Oak, Michigan
  - Ascension Providence Hospital, Southfield, Michigan
  - Gates Vascular Institute / SUNY Buffalo, Buffalo, New York
  - Lenox Hill Hospital / Northwell Health, New York, New York
  - OhioHealth Riverside, Columbus, Ohio
  - Penn Presbyterian/Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Lankenau Medical Center / Pulmonology Associates, Wynnewood, Pennsylvania
  - Inova Fairfax, Falls Church, Virginia

REFERENCES:
- [Result] Silver MJ, Gibson CM, Giri J, Khandhar S, Jaber W, Toma C, Mina B, Bowers T, Greenspon L, Kado H, Zlotnick DM, Chakravarthy M, DuCoffe AR, Butros P, Horowitz JM. Outcomes in High-Risk Pulmonary Embolism Patients Undergoing FlowTriever Mechanical Thrombectomy or Other Contemporary Therapies: Results From the FLAME Study. Circ Cardiovasc Interv. 2023 Oct;16(10):e013406. doi: 10.1161/CIRCINTERVENTIONS.123.013406. Epub 2023 Oct 17. PMID 37847768
- See also: Outcomes in High-Risk Pulmonary Embolism Patients Undergoing FlowTriever Mechanical Thrombectomy or Other Contemporary Therapies: Results From the FLAME Study — https://pubmed.ncbi.nlm.nih.gov/37847768/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients presenting to the hospital/emergency department with PE or who incidentally develop PE while in the hospital were assessed for high-risk PE, and for eligibility for enrollment in the FLAME study.
Pre-assignment Details: Subjects who met eligibility criteria for the study and had a primary thrombus removal strategy initiated were enrolled into either the FlowTriever, Context or Prior Therapy Arm, based on the thrombus removal strategy initiated. These three arms were non-randomized parallel registries.
Groups:
- FlowTriever Arm: Subjects treated with FlowTriever thrombectomy as the primary treatment strategy for high-risk PE
- Context Arm: Subjects treated with any other approach as the primary treatment strategy for high-risk PE (including non-FlowTriever mechanical thrombectomy [0%], anticoagulation alone [23.0%] systemic thrombolysis [68.9%], catheter-directed thrombolysis [6.6%], or surgical thrombectomy [1.6%]
- Prior Therapy Arm: Subjects presenting with low or intermediate-risk PE who received advanced therapy but subsequently progressed to high-risk PE in the same hospital setting/admission
Period: Overall Study
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
Started | 53 | 61 | 1
Completed | 48 | 43 | 0
Not Completed | 5 | 18 | 1
Not completed — Death | 1 | 18 | 1
Not completed — Remained in-hospital for >/= 45 Days | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Context Arm: Subjects treated with any other approach as the primary treatment strategy for high-risk PE (including non-FlowTriever mechanical thrombectomy [0%], anticoagulation alone [23.0%], systemic thrombolysis [68.9%], catheter-directed thrombolysis [6.6%], or surgical thrombectomy [1.6%])
- Prior Therapy Arm: Subjects presenting with low- or intermediate-risk PE who received advanced therapy but subsequently progressed to high-risk PE in the same hospital setting/admission
- Total: Total of all reporting groups
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm | Total
Number analyzed (Participants) | 53 | 61 | 1 | 115
Age, Continuous [Mean (Full Range); unit: years] | 64.8 [26 to 92] | 61.6 [33 to 89] | 58.0 [58 to 58] | 63.0 [26 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 35 | 1 | 62
  Male | 27 | 26 | 0 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 39 | 43 | 0 | 82
  Unknown or Not Reported | 13 | 16 | 1 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Of the "Unknown or Not Reported" Races; 4 were not provided in FlowTriever Arm, 2 were not provided in the Context Arm, and 1 was not provided in the Prior Therapy Arm. Additionally, 1 Context Arm Race was reported as "Other"
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 16 | 40 | 0 | 56
    White | 33 | 18 | 0 | 51
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 4 | 3 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 53 | 61 | 1 | 115

OUTCOME MEASURES:

1. Primary Outcome: Composite Incidence of All-cause Mortality, Clinical Deterioration, Bailout, and Major Bleeding
Description: The primary endpoint is the in-hospital composite endpoint of all-cause mortality, bailout to an alternative thrombus removal strategy, clinical deterioration, and major bleeding (BARC 3b/3c/5a/5b definition). The primary endpoint was assessed in the FlowTriever Arm compared to a pre-specified performance goal of 32%.
  Subjects in the Context Arm were analyzed separately using descriptive methods. The primary endpoint in the Context Arm was not compared to a performance goal. Data collection for Prior Therapy Arm subjects included information surrounding the PE treatment, progression to High-Risk PE, and patient course through hospital discharge. Safety data were collected, but not CEC adjudicated or analyzed as outlined for the FlowTriever and Context Arm subjects.
Time Frame: From the time of primary treatment for high-risk pulmonary embolism through hospital discharge or 45 days, whichever comes first.
Population: All patients in the FlowTriever Arm and Context Arm. Data collection for Prior Therapy Arm subjects included information surrounding the PE treatment, progression to High-Risk PE, and patient course through hospital discharge. Safety data were collected, but not CEC adjudicated or analyzed as outlined for the FlowTriever and Context Arm subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 9 | 39

2. Secondary Outcome: All-Cause Mortality
Description: Incidence of mortality
Time Frame: as for outcome 1
Population: All patients in the FlowTriever Arm and Context Arm. Safety data were collected, but not CEC adjudicated or analyzed as outlined for the FlowTriever and Context Arm subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 1 | 18

3. Secondary Outcome: Bailout to an Alternative Thrombus Removal Strategy
Description: Incidence of bailout to an alternative thrombus removal strategy
Time Frame: as for outcome 1
Population: All patients in the FlowTriever and Context Arm. Safety data were collected, but not CEC adjudicated or analyzed as outlined for the FlowTriever and Context Arm subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 2 | 16

4. Secondary Outcome: Clinical Deterioration
Description: Incidence of clinical deterioration
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 8 | 13

5. Secondary Outcome: Major Bleeding
Description: Incidence of major bleeding
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 6 | 15

6. Secondary Outcome: Frequency of Stroke
Description: Incidence of ischemic or hemorrhagic stroke
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 1 | 4

7. Secondary Outcome: Device-related Complications
Description: Incidence of device-related complications
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 12 | 10

8. Secondary Outcome: Access Site Injury Requiring Intervention, Both Venous and Arterial
Description: Incidence of access site injury requiring intervention, including both venous and arterial
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm
Number analyzed (Participants) | 53 | 61
Participants | 4 | 5

9. Other Pre Specified Outcome: Length of Hospital Stay
Description: Length of post-treatment hospital stay, measured in number of overnights
Time Frame: as for outcome 1
Population: All patients in FlowTriever, Context and Prior Therapy Arms who survived to discharge or 45 days, whichever comes first.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Prior Therapy Arm: Subjects presenting with low- or intermediate-risk PE who received advanced therapy but subsequently processed to high-risk PE in the same hospital setting/admission
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
Number analyzed (Participants) | 52 | 43 | 0
Days | 7 [3 to 12.5] | 8 [6 to 15] |

10. Other Pre Specified Outcome: Length of ICU Stay
Description: Length of post-treatment ICU stay, measure in number of overnights
Time Frame: From treatment start or ICU admission, whichever is later, to ICU discharge
Population: All patients in the FlowTriever, Context and Prior Therapy Arms who survived to discharge or study exit
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
Number analyzed (Participants) | 52 | 43 | 0
Days | 2 [1 to 4] | 3 [1 to 7] |

11. Other Pre Specified Outcome: Use of ECMO
Description: Frequency of ECMO use, including either pre or post treatment initiation
Time Frame: as for outcome 1
Population: All patients in FlowTriever, Context and Prior Therapy Arms
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
Number analyzed (Participants) | 53 | 61 | 1
Participants | 3 | 7 | 0

12. Other Pre Specified Outcome: Discharge Location
Description: Discharge location after hospital stay
Time Frame: as for outcome 1
Population: All patients in the FlowTriever, Context and Prior Therapy Arms
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
Number analyzed (Participants) | 53 | 61 | 1
Participants
  Home | 26 | 23 | 0
  Home with healthcare | 6 | 3 | 0
  Care facility/skilled nursing home | 13 | 11 | 0
  Stayed in hospital for >/= 45 days | 4 | 0 | 0
  Expired prior to discharge | 1 | 18 | 1
  Other | 3 | 6 | 0

13. Other Pre Specified Outcome: Time to Extubation
Description: Time to extubation reported as number of days
Time Frame: From the time of initiation of primary treatment to extubation
Population: All patients in the FlowTriever Arm, Context Arm and Prior Therapy arm who survived to discharge or study exit, underwent a single intubation procedure prior to initiation of primary treatment, and were extubated prior to and through discharge or study exit
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
Number analyzed (Participants) | 4 | 6 | 0
Days | 1.640 [1.200 to 4.305] | 1.795 [1.530 to 3.060] |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of enrollment through hospital discharge (or through day 45, whichever occurred first)
Description: The study only captured AEs related to the subject's PE condition and treatment. Reportable AEs included all events considered in the safety analyses, all thrombus removal therapy/device- and/or procedure-related AEs, as well as events resulting in death. For the Prior Therapy arm, safety data were collected but not CEC adjudicated or analyzed.
Arm/Group | FlowTriever Arm | Context Arm | Prior Therapy Arm
All-Cause Mortality (participants affected / at risk) | 1/53 | 18/61 | 1/1
Serious Adverse Events (participants affected / at risk) | 16/53 | 37/61 | 1/1
Other Adverse Events (participants affected / at risk) | 10/53 | 19/61 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FlowTriever Arm (N=53) | Context Arm (N=61) | Prior Therapy Arm (N=1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Brain Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Breast haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Chest wall haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orbital haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
Pulmonary haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 8 (8) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth socket haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0)
Worsening Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Worsening Shock Liver (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FlowTriever Arm (N=53) | Context Arm (N=61) | Prior Therapy Arm (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue biting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tongue haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04795167/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04795167/SAP_001.pdf